CLINICAL TRIAL: NCT01762007
Title: The Change of the Detrusor Thickness After Hypospadias Repair - Comparison With the Normal Control Group
Status: Withdrawn | Type: Observational
Why Stopped: Due to difficulty in purchasing reagents, study canceled without subject registration
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2012-0372
Record Dates: First submitted 2012-12-19; First posted 2013-01-07 (Estimated); Last update posted 2021-05-06 (Actual); Status verified 2021-05

CONDITIONS: Hypospadias
Keywords: hypospadias, bladder outlet obstruction, ultrasonography
MeSH Terms: conditions — Hypospadias; Urinary Bladder Neck Obstruction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- 6Mo-2Yr old penile hypospadias patients before operation
- 6Mo-2Yr old male patients without hypospadias
- penile hypospadias patients under the age of 5 Yr: penile hypospadias patients under the age of 5 Yr who got tubularized incised plate operation at out institution at the age between 6Mo and 2Yr old and more than 1 Yr have passed
- 2Yr-5Yr old male patients without hypospadias

SUMMARY:
Even successfully managed hypospadias without any complication, voiding problem could be developed due to the increased urethral resistance. The investigators are trying to analyze the effect of hypospadias operation on voiding function by checking the detrusor thickness and urinary nerve growth factor.

ELIGIBILITY:
Inclusion Criteria:

<Group 1>

1. 6Mo-2Yr old penile hypospadias patients before operation <Group 2>
2. 6Mo-2Yr old male patients without hypospadias <Group 3>
3. penile hypospadias patients under the age of 5 Yr who got tubularized incised plate operation at out institution at the age between 6Mo and 2Yr old and more than 1 Yr have passed <Group 4>
4. 2Yr-5Yr old male patients without hypospadias1. 0-3 year old children without any abnormality of urinary tract

Exclusion Criteria:

<Group 1, 2, 4>

1. patients with history of urethral operation, febrile urinary tract infection, neurogenic abnormality om operation <Group 3>

1. patients with history of urethral operation other than hypospadias repair, febrile urinary tract infection, neurogenic abnormality
2. patients with development urethra-cutaneous fistula

Max Age: 5 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Group 1: 13 patients with 6Mo-2Yr old penile hypospadias patients before operation Group 2: 13 patients with 6Mo-2Yr old male patients without hypospadias Group 3: 15 patients with penile hypospadias patients under the age of 5 Yr who got tubularized incised plate operation at out institution at the age between 6Mo and 2Yr old and more than 1 Yr have passed Group 4: 15 patients with 2Yr-5Yr old male patients without hypospadias
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2012-11; Primary Completion 2013-07 (Estimated); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
Detrusor thickness | immediate analysis of detrusor thickness at the enrollment time of this study

SECONDARY OUTCOMES:
urinary nerve growth factor level | immediate analysis of urinary nerve growth factor level at the enrollment time of this study

CONTACTS AND LOCATIONS:
Locations (1):
- Sang Won, Seoul, South Korea